CLINICAL TRIAL: NCT06675045
Title: Description of Respiratory Variability in Patients With Acute Hypoxemic Respiratory Failure and Placed on High Flow Oxygen Therapy - Exploratory Study
Brief Title: Respiratory Variability in Patients With Acute Hypoxemic Respiratory Failure and Placed on High Flow Oxygen Therapy
Acronym: HYPOXEVARIA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-A01080-47
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Acute Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Respiratory Variability Monitoring (Experimental): Respiratory variability will be measured using a belt equipped with an external sensor allowing automatic and continuous analysis of thoracic movement by frequency analysis
  Interventions: Other: Respiratory variability monitoring

INTERVENTIONS:
Other: Respiratory variability monitoring — Respiratory variability will be measured using a belt equipped with an external sensor allowing automatic and continuous analysis of thoracic movement by frequency analysis

SUMMARY:
Recommendations from the European Respiratory Society are to use high-flow oxygen therapy rather than conventional oxygen therapy and non-invasive ventilation (NIV) in cases of acute hypoxaemic respiratory failure.

Studies have shown that high-flow oxygen therapy can reduce the need for intubation and the initiation of NIV without reducing mortality. In addition, by improving oxygenation, high-flow oxygen therapy can create a feeling of security which may delay endotracheal intubation.

Two studies have suggested that mortality is higher in patients receiving delayed intubation (≥ 48 hours) after failure of high flow oxygen therapy. Another study suggests that delayed endotracheal intubation after high-flow oxygen therapy ≥ 48 hours increases the risk of patient mortality independently of comorbidities and severity of illness on admission. Finally, other results suggest that the increased risk of mortality may be significant after 36 hours of high-flow oxygen therapy. It is therefore difficult to determine the right time for intubation and invasive ventilation.

A diagnostic decision aid could be of great use to the attending physician in optimising the patient's respiratory assistance strategy, whether invasive or non-invasive. Consequently, any clinical marker that can provide early detection of altered respiratory status on high-flow oxygen therapy deserves to be evaluated.

Respiratory variability is synonymous with respiratory 'good health'. A decrease in this same variabilitý is pathological and indicates an increase in the level of loads imposed on the respiratory system. It means that the measurement of respiratory variability indices may be one of these markers

There are devices for non-invasive, continuous monitoring of respiratory variability, with automated frequency analysis of thoracic movement. In this study, respiratory variability indices will be measured in patients admitted to intensive care under high-flow oxygen therapy using an external sensor called REVAMODE.

DETAILED DESCRIPTION:
Recommendations from the European Respiratory Society are to use high-flow oxygen therapy rather than conventional oxygen therapy and non-invasive ventilation (NIV) in cases of acute hypoxaemic respiratory failure.

Studies have shown that high-flow oxygen therapy can reduce the need for intubation and the initiation of NIV without reducing mortality. In addition, by improving oxygenation, high-flow oxygen therapy can create a feeling of security which may delay endotracheal intubation. Delaying intubation would expose the patient to respiratory effort, leading to self-inflicted lung injury by a mechanism similar to ventilation-induced lung injury. Self-inflicted lung injury may increase mortality in acute respiratory distress syndrome (ARDS).

Two studies have suggested that mortality is higher in patients receiving delayed intubation (≥ 48 hours) after failure of high flow oxygen therapy. Another study suggests that delayed endotracheal intubation after high-flow oxygen therapy ≥ 48 hours increases the risk of patient mortality independently of comorbidities and severity of illness on admission. Finally, other results suggest that the increased risk of mortality may be significant after 36 hours of high-flow oxygen therapy. It is therefore difficult to determine the right time for intubation and invasive ventilation.

A diagnostic decision aid could be of great use to the attending physician in optimising the patient's respiratory assistance strategy, whether invasive or non-invasive. Consequently, any clinical marker that can provide early detection of altered respiratory status on high-flow oxygen therapy deserves to be evaluated.

Respiratory variability is synonymous with respiratory 'good health'. A decrease in this same variabilitý is pathological and indicates an increase in the level of loads imposed on the respiratory system. For this reason, this study is based on the hypothesis that the measurement of respiratory variability indices may be one of these markers.

There are devices for non-invasive, continuous monitoring of respiratory variability, with automated frequency analysis of thoracic movement. In this study, respiratory variability indices will be measured in patients admitted to intensive care under high-flow oxygen therapy using an external sensor called REVAMODE.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, aged ≥ 18 years
* Patient admitted to intensive care with acute hypoxaemic respiratory failure
* Patient treated with high-flow oxygen therapy

Exclusion Criteria:

* Patient admitted to intensive care with invasive ventilation
* Patient with therapeutic abstention for intubation
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Coefficient of variation | Day 1 and Day 2
  Each respiratory cycle is defined by an inspiratory time followed by an expiratory time.

CONTACTS AND LOCATIONS:
Overall Officials: Kais BEN HASSEN, MD, Principal Investigator — Hôpital privé de Clairval

IPD SHARING:
Plan to Share IPD: No